CLINICAL TRIAL: NCT06280716
Title: A Multicenter, Randomized, Double-Blind, Placebo-controlled, Phase 3 Trial to Investigate the Efficacy and Safety of Lebrikizumab When Used With/Without Topical Corticosteroid Treatment in Participants With Moderate-To-Severe Atopic Dermatitis
Brief Title: A Study of Lebrikizumab (LY3650150) With/Without Topical Corticosteroid Treatment in Participants With Moderate-to-Severe Atopic Dermatitis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18817; J2T-MC-KGBW (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — lebrikizumab; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel group, placebo controlled
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Lebrikizumab every 2 weeks (Q2W) (Experimental): Induction Period (Baseline-Week 16):
  Two subcutaneous (SC) injections of lebrikizumab as a loading dose at Baseline and Week 2 followed by a single injection every 2 weeks (Q2W) from Week 4 until Week 14. Induction period includes mono cohort with only lebrikizumab and combo cohort where lebrikizumab is in combination with TCS treatment.
  Interventions: Drug: Lebrikizumab; Drug: Topical Corticosteroid
- Lebrikizumab every 4 weeks (Q4W) (Experimental): Maintenance Period (Week 16-Week 52):
  Treatment from Week 16 to Week 52 is based on re-randomization of responders (from lebrikizumab Q2W arm) in the Induction Period. Participants re-randomized to the Lebrikizumab Q4W arm receive one lebrikizumab injection Q4W from Week 16 until Week 48.
  Interventions: Drug: Lebrikizumab
- Lebrikizumab every 8 weeks (Q8W) (Experimental): Maintenance Period (Week 16-Week 52):
  Treatment from Week 16 to Week 52 is based on re-randomization of responders (from lebrikizumab Q2W arm) in the Induction Period. Participants re-randomized to Lebrikizumab Q8W arm receive one lebrikizumab injection Q8W, with one placebo injection 4 weeks after each lebrikizumab injection from Week 16 until Week 48.
  Interventions: Drug: Lebrikizumab
- Escape Arm (Lebrikizumab Q2W) (Experimental): Maintenance Period (Week 16-Week 50):
  Participants who require rescue treatment for atopic dermatitis (AD) during the Induction Period, or are non-responders at Week 16, will be eligible for treatment in an Escape Arm where participants will receive open label lebrikizumab Q2W from Week 16 through Week 50. In addition, participants who do not maintain an acceptable response during the Maintenance Period (have an EASI score <50% of baseline), will be eligible for the Escape Arm.
  Interventions: Drug: Lebrikizumab
- Placebo (Placebo Comparator): Induction Period (Baseline-Week 16):
  Two subcutaneous (SC) injections of Placebo as a loading dose at Baseline and Week 2 followed by a single injection every 2 weeks (Q2W) from Week 4 until Week 14. Induction period includes mono cohort with only Placebo and combo cohort where Placebo is given in combination with topical corticosteroid (TCS) treatment.
  Maintenance Period (Week 16-Week 52):
  Participants of responders at Week 16 will receive single injection of placebo every 4 weeks (Q4W) from Week 16 until Week 48.
  Interventions: Drug: Placebo; Drug: Topical Corticosteroid

INTERVENTIONS:
Drug: Placebo — Subcutaneous injection
  Arms: Placebo
Drug: Lebrikizumab — Subcutaneous injection
  Other Names: LY3650150
  Arms: Escape Arm (Lebrikizumab Q2W); Lebrikizumab every 2 weeks (Q2W); Lebrikizumab every 4 weeks (Q4W); Lebrikizumab every 8 weeks (Q8W)
Drug: Topical Corticosteroid — Topical Corticosteroid
  Arms: Lebrikizumab every 2 weeks (Q2W); Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of lebrikizumab with/without Topical Corticosteroid Treatment in Participants with Moderate-to-Severe Atopic Dermatitis. The study will last approximately 62 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic AD that has been present for ≥1 year before the screening period or have chronic eczema and meet the AAD criteria.
* Have moderate-to-severe AD, including all of the following at the baseline: EASI score ≥16, IGA score ≥3 (scale of 0 to 4), ≥10% BSA of AD involvement.
* Have a documented history provided by a physician and/or investigator of inadequate response to existing topical medications within 6 months preceding screening as defined by at least 1 of the following:

  1. Inability to achieve good disease control, defined as mild disease or better after use of at least a medium-potency TCS for at least 4 weeks, or for the maximum duration recommended by the product prescribing information, whichever is shorter. TCS may be used with or without TCIs and/or topical Janus kinase (JAK) inhibitors.
  2. Participants who failed systemic therapies intended to treat AD within 6 months preceding screening, such as cyclosporine, MTX, azathioprine, and MMF, will also be considered as surrogates for having inadequate response to topical therapy.
* Adolescents body weight must be ≥40 kg at baseline.
* Males may participate in this trial and comply with specific local government study requirements. Females of childbearing potential and females not of childbearing potential may participate in this trial.

Exclusion Criteria:

* Have received a dose of lebrikizumab in any prior lebrikizumab clinical study.
* Have a history of anaphylaxis or uncontrolled chronic disease that might require bursts of oral corticosteroids.
* Have a current or recent acute, active infection. For at least 30 days before screening and up to the randomization, participants must have no symptoms or signs of confirmed or suspected infection and must have completed any appropriate anti-infective treatment.
* Have had Serious, Opportunistic, Chronic and Recurring infection within 3 months prior to the screening or develops any of these infections before the randomization.
* Have active tuberculosis (TB) or latent tuberculosis infection (LTBI) that has not been treated with a complete course of appropriate therapy or such treatment is underway.
* Have a current infection with HBV, HCV, human immunodeficiency virus (HIV) infection.
* Have presence of skin comorbidities that may interfere with study assessments.
* Have a diagnosis or history of malignant disease within 5 years before screening, with the following exceptions:

  1. basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years, and
  2. cervical carcinoma in situ, with no evidence of recurrence within 5 years before screening visit.
* Pregnant or breastfeeding women or women planning to become pregnant or breastfeed during the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Eczema Area and Severity Index (EASI-75) (≥75% Reduction in EASI Score) for Mono Cohort | Week 16
  The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent, i.e., percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 (none) to 72 (severe).
  The EASI-75 responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the EASI score
Percentage of Participants Achieving EASI-75 for Combo Cohort | Week 16
  The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent, i.e., percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI-75 score was obtained by weight-averaging these 4 scores and will range from 0 (none) to 72 (severe).
  The EASI-75 responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the EASI score.
Percentage of Participants Achieving IGA Score of 0 or 1 and a Reduction of ≥2 Points From Baseline to Week 16 for Mono Cohort | Baseline, Week 16
  The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Percentage of Participants Achieving IGA Score of 0 or 1 and a Reduction of ≥2 Points From Baseline to Week 16 for Combo Cohort | Baseline, Week 16
  The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification. when used in combination with TCS treatment.

SECONDARY OUTCOMES:
Percentage of Participants Achieving EASI-90 (≥90% Reduction in EASI Score) for Combo Cohort | Week 16
  The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent, i.e., percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 (none) to 72 (severe).
  The EASI-90 responder is defined as a participant who achieves a ≥ 90% improvement from baseline in the EASI score.
Percentage of Participants With a Itch Numerical Rating Scale (NRS) Score of ≥4-Points at Baseline who Achieve a ≥4-Point Reduction in Itch NRS Score From Baseline to Week 16 for Combo Cohort | Baseline, Week 16
  Itch NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours with 0 indicating "No itch" and 10 indicating "Worst itch imaginable."
Percentage Change From Baseline in EASI Score for Combo Cohort | Baseline, Week 16
  The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease, i.e., percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 (none) to 72 (severe).
Percent Change from Baseline in Itch Numeric Rating Scale (NRS) for Combo Cohort | Baseline, Week 16
  The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable". Overall severity of a participant's itching is indicated by selecting the number that best describes the worst level of itching in the past 24 hours (Naegeli et al. 2015; Kimball et al. 2016; Newton et al. 2019; Silverberg et al. 2021). The Itch NRS assessment will be completed daily by the participant using a handheld device.
Change from Baseline in Dermatology Life Quality Index (DLQI) for Combo Cohort | Baseline, Week 16
  The DLQI is a participant-reported, 10-item, quality-of-life questionnaire in those ≥16 years of age that covers 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment). The recall period of this scale is over the "last week." Response categories include "not at all," "a little", "a lot," and "very much," with corresponding scores of 0, 1, 2, and 3, respectively, and unanswered (or "not relevant") responses scored as 0.
  Scores range from 0 to 30 with higher scores indicating greater impairment of QoL. A DLQI total score of 0 to 1 is considered as having no effect on a participant's health related quality-of-life (HRQoL), and a 4-point change from baseline is considered as the minimal clinically important difference threshold.
Percentage of Participants Achieving EASI-90 for Mono Cohort | Week 16
  The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent, i.e., percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 (none) to 72 (severe).
  The EASI-90 responder is defined as a participant who achieves a ≥ 90% improvement from baseline in the EASI score
Percentage of Participants With a Itch NRS Score of ≥4-Points at Baseline who Achieve a ≥4-Point Reduction in Itch NRS Score From Baseline to Week 16 for Mono Cohort | Baseline, Week 16
  Itch NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours with 0 indicating "No itch" and 10 indicating "Worst itch imaginable."
Percentage Change From Baseline in EASI Score for Mono Cohort | Week 16
  The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease, i.e., percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 (none) to 72 (severe).
Percent Change from Baseline in Itch Numeric Rating Scale (NRS) for Mono Cohort | Baseline, Week 16
  The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable". Overall severity of a participant's itching is indicated by selecting the number that best describes the worst level of itching in the past 24 hours (Naegeli et al. 2015; Kimball et al. 2016; Newton et al. 2019; Silverberg et al. 2021). The Itch NRS assessment will be completed daily by the participant using a handheld device
Change from Baseline in Dermatology Life Quality Index (DLQI) for Mono Cohort | Baseline, Week 16
  The DLQI is a participant-reported, 10-item, quality-of-life questionnaire in those ≥16 years of age that covers 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment). The recall period of this scale is over the "last week." Response categories include "not at all," "a little", "a lot," and "very much," with corresponding scores of 0, 1, 2, and 3, respectively, and unanswered (or "not relevant") responses scored as 0.
  Scores range from 0 to 30 with higher scores indicating greater impairment of QoL. A DLQI total score of 0 to 1 is considered as having no effect on a participant's health related quality-of-life (HRQoL), and a 4-point change from baseline is considered as the minimal clinically important difference threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (46):
- China (41):
  - Wannan Medical College Yijishan Hospital, Wuhu, Anhui
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Children's hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Affiliate of Capital University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - The Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Zhongshan Hospital Fudan University (Xiamen Branch), Xiamen, Fujian
  - Guangdong Province Dermatology Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Hospital of Wuhan, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi No.2 People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Children's Hospital of Shanxi, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First People's Hospital of Hangzhou, Hangzhou, Zhejiang
  - The first Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang University School of Medicine - The Fourth Affiliated Hospital, Yiwu, Zhejiang
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou
  - Shanghai Skin Disease Hospital, Shanghai
- South Korea (5):
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Bupyeong-gu, Incheon-gwangyeoksi [Incheon]
  - Korea University Ansan Hospital, Ansan-si, Kyǒnggi-do
  - National Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Hallym University Kangnam Sacred Heart Hospital, Seoul, Seoul-teukbyeolsi [Seoul]

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement
URL: http://vivli.org/

REFERENCES:
- See also: Related Info — https://trials.lilly.com/en-US/trial/464995